CLINICAL TRIAL: NCT01113281
Title: Phase Ib Open Label, Randomized, Controlled, Dose-Escalation Study to Evaluate Safety and Immunogenicity of VPM1002 in Comparison With BCG in Healthy Volunteers in South Africa
Brief Title: Dose-Escalation Study on Safety and Immunogenicity of VPM1002 in Comparison to BCG in Healthy Volunteers in South Africa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Serum Life Science Europe GmbH (Industry)
Collaborators: Farmovs-Parexel Bloemfontein, Republic of South Africa (Clinical Site) (Unknown); Triclinium Johannesburg, RSA (Monitoring and Overall Management of the study) (Unknown); University of Stellenbosch (Other); HJ-CTC George, RSA (Statistics & Report) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VPM1002-ZA-1.10TB; DOH-27-0210-3083 (Other: NHREC (National Health Researh Ethics Council) South Africa)
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine; Live Vaccine; rBCG
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VPM1002 in three dosages (Experimental)
  Interventions: Biological: VPM1002 live vaccine
- BCG (Active Comparator)
  Interventions: Biological: commercially available live vaccine BCG

INTERVENTIONS:
Biological: VPM1002 live vaccine
  Arms: VPM1002 in three dosages
Biological: commercially available live vaccine BCG
  Arms: BCG

SUMMARY:
Goal of VPM is the development of a recombinant urease C-deficient listeriolysin expressing BCG vaccine strain (VPM1002) as a safe, well tolerated and efficacious vaccine against tuberculosis (TB) for residents in endemic areas and persons at risk in non-endemic areas. The new vaccine should be at least as potent as the current strain and should be safer than BCG (Kaufmann, 2007a; Grode et al., 2005). The vaccine is formulated as live lyophilised bacteria to be re-suspended before intradermal injection. The preceding clinical trial in 80 volunteers in Germany indicated immunogenicity and safety being sufficient for proceeding with the clinical development. Hence, the current study is commenced in South Africa, a country highly endemic for tuberculosis.

24 volunteers were randomly allocated to 4 groups each with 6 adult healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers 18 to 45 years of age
* Volunteers must use acceptable contraception and avoid pregnancy for the duration of the study (6 months)
* Healthy (medical history, physical examination, vital signs, ECG and laboratory tests at screening)
* No signs of active or latent tuberculosis infection
* BMI of 19 - 33 kg/m2
* Subjects must be able and willing to comply with the study protocol, available and willing to complete all study measurements and have signed an Informed Consent form approved by the Ethics Committee.
* Reachable by phone during the whole study period (approximately 6 months).
* Negative test for HIV1 and HIV2, hepatitis B surface antigen and antibody to hepatitis C virus.
* No anamnestic evidence for a primary or secondary immunodeficiency.
* No skin eczema lesion at the intended injection site.
* No anamnestic predisposition for scarring badly or for keloid formation.
* No other vaccination during eight weeks before the current study.
* No participation in another clinical trial within 3 months before study vaccination and the 6 months of the current study.
* No prior participation in a TB vaccine trial.
* Able and willing to abstain from strenuous physical exercise 24 hours before screening examination, and 24 hours before vaccination

Exclusion Criteria:

* History of prior TB disease
* History of anaphylaxis or severe allergic reactions
* Known allergies to any component of the investigational or reference product or known history of severe skin reaction against the Tuberculin test
* Presence of any person in the household of the volunteer with active tuberculosis disease
* Tuberculin-PPD-in-vivo-test equal or more than 10 mm before baseline
* systemic disorders which could interfere with the interpretation of the study results or compromise the health of the volunteers
* BCG-vaccination during 10 years before study vaccination
* Acute fever or fever in the last 7 days before dosing
* Any malignant condition
* Concomitant treatment with medication that may affect immune function during 3 months before study vaccination and the 6 months of current study. No oral antibiotics during the 14 days before study vaccination and no injectable antibiotics during the 28 days prior to vaccination.
* Treatment with blood products in the past 6 months up to end of study.
* Any clinically significant laboratory abnormalities on screened blood samples.
* A history of drug or alcohol abuse
* Positive test for drugs of abuse on urine testing at screening
* Blood donation for non study-related purposes within 3 months before and during the entire duration of the study
* Clinically relevant result from sonographic liver imaging
* Professional or regular contact with live animals for food production

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Safety: physical examination, vital signs, electrocardiogram, liver sonography, laboratory safety parameters, tolerability, recording of concomitant medication and adverse events | baseline, days 2, 7, 14, 28, 56, and month 6

SECONDARY OUTCOMES:
Immunogenicity: Interferon-gamma-ELISA (IFN-g-ELISA) in supernatants of peripheral blood mononuclear cells (PBMC) restimulated with tuberculin (PPD from Staten Serum Institute, Denmark) | baseline, days 14, 28, 56 and month 6
Immunogenicity: ELISPOT for the number of IFN-g-secreting PBMC after restimulation with PPD | baseline, days 14, 28, 56 and month 6
Immunogenicity: Whole Blood Assays (WBA): IFN-g-ELISA of supernatants of whole blood restimulated with PPD | baseline, days 14, 28, 56 and month 6
Immunogenicity: Intracellular Cytokine Staining (ICS) for IFN-g, TNF-a and IL-2 in CD4+ and CD8+ lymphocytes upon stimulation with PPD | baseline, days 14, 28, 56 and month 6
Immunogenicity: ICS with other triple combinations of markers in CD4+ and CD8+ lymphocytes upon stimulation with PPD | baseline, days 14, 28, 56 and month 6
Immunogenicity: Antigen-85B (Ag85B) and BCG as recall antigens for ELISA, ELISPOT, WBA and ICS | baseline, days 14, 28, 56 and month 6
Immunogenicity: serum antibodies against PPD or Ag85B | baseline, days 14, 28, 56 and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Mada Ferreira, MD, Principal Investigator — Farmovs-Parexel, Bloemfontein, RSA
Locations (1):
- Farmovs-Parexel, Bloemfontein, South Africa